CLINICAL TRIAL: NCT02410057
Title: ALFoNS - Growth and Metabolism in Infants Fed Protein-reduced, Alpha-lactalbumin Enriched Formula Compared to Breastfed Infants
Brief Title: Growth and Metabolism in Infants Fed Protein-reduced, Alpha-lactalbumin Enriched Formula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Skane University Hospital (Other)
Collaborators: University of California, Davis (Other); Umeå University (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Pia Karlsland Åkeson, MD, PhD, Senior Consultant, Lund University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SkaneUH
Record Dates: First submitted 2015-03-20; First posted 2015-04-07 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Growth; Infection; Sleep
Keywords: growth; formula; protein; alpha-lactalbumin; amino acids; metabolomics; microbiota
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard infant formula (Active Comparator): Standard infant formula
  Interventions: Dietary Supplement: Standard infant formula
- Protein-reduced whey formula (Experimental): Protein-reduced whey formula with higher level of α-lactalbumin than in standard infant formula
  Interventions: Dietary Supplement: Protein-reduced whey formula
- Protein-reduced α-lactalbumin formula (Experimental): Protein-reduced formula with level of α-lactalbumin more similar to breast milk and higher than in experimental whey formula and in standard infant formula
  Interventions: Dietary Supplement: Protein-reduced α-lactalbumin formula
- Breast-feeding (No Intervention): Exclusive breast-feeding

INTERVENTIONS:
Dietary Supplement: Protein-reduced α-lactalbumin formula — Protein-reduced formula with levels of α-lactalbumin more similar to breast milk and higher than in whey formula and in standard infant formula
  Arms: Protein-reduced α-lactalbumin formula
Dietary Supplement: Protein-reduced whey formula — Protein-reduced whey formula with higher levels of α-lactalbumin than in standard infant formula
  Arms: Protein-reduced whey formula
Dietary Supplement: Standard infant formula — Standard infant formula
  Arms: Standard infant formula

SUMMARY:
Formula composition is developed to resemble breast milk as close as possible, but there are still considerable differences between formula and breast milk composition, probably resulting in higher risk of overweight in childhood and higher incidence of infections in formula-fed infants. Protein levels are still higher and constituents such as alpha-lactalbumin lower in formula than in breast milk. By adding more alpha-lactalbumin to formula, rich in tryptophan, the resulting amino acid composition will allow further reduction of protein in formula. The investigators intend to include 320 infants, where 80 will be exclusively breastfed and the remainder assigned in a double blind, controlled, randomized manner to one of three formula groups; two experimental, protein reduced formula with two different levels of alpha-lactalbumin and one group given standard infant formula. The intervention period is from 4-8 weeks until 6 months of age. The infants will be followed by growth parameters, blood-, urine- and fecal biomarkers and health parameters until 5 years of age. The experimental formula will possibly result in growth, metabolism and gut microbiota as well as health parameters more similar to those of breastfed infants

DETAILED DESCRIPTION:
Background: Breast milk is the best source of nutrition for the rapidly growing infant since it contains all the necessary nutrients in the right proportions. If the mother cannot breast-feed, chooses not to breast-feed or has to stop early, an adapted formula is from a nutritional perspective the only alternative during the first four to six months of age and also the best alternative throughout the rest of the first year of life together with suitable complementary foods. Formula composition has through the years developed to resemble as close as possible the composition of breast milk resulting in physiological effects in the infant to more resemble that of the breast-fed infant. However, there are still considerable differences between the dietary intake of the breast-fed infant and its metabolism compared to infants who are fed formula. Furthermore, research suggests that breast-fed infants have a lower risk of overweight and obesity in childhood and adolescence, lower risk of acute otitis media (AOM), upper airway- and gastrointestinal infections, and possibly a lower risk of high blood pressure and diabetes type 2 as adults which probably depend on different protein composition and concentration in formula and breastmilk. The optimal protein level of formula is still under debate. The investigators know that the protein concentration of formula is unnecessarily high, but until now it has been difficult to reduce it further due to the potential risk of shortage of some of the essential amino acids, i.e. those amino acids that have to be delivered from the diet.

The concentration of alpha-lactalbumin, the predominating whey protein in breast milk, is still low in formula. The composition of the protein in breast milk and formula thus differs considerably and consequently also the amino acid pattern in serum between infants who are breast-, or formula-fed. Alpha-lactalbumin has many potential positive effects which may explain some of the differences between breast-fed and formula-fed infants and when added to formula makes it more similar to the composition of breast milk. Alpha-lactalbumin contains a higher concentration of cysteine, a precursor of taurine, which is important for neurodevelopment. However, it is foremost the concentration of tryptophan that is higher in alpha-lactalbumin, an amino acid which otherwise is a limiting factor when lowering the protein level in formula. Tryptophan is a precursor of serotonin, a neurotransmitter important for stress management, cognition under stress and sleep latency.

Recently, new whey protein sources which contain higher concentrations of alpha-lactalbumin have become available. Studies show that protein is still too high in formula resulting in higher concentrations of urea nitrogen and most amino acids in infants who are fed formula compared to those who are breast-fed, which indicates that formula-fed infants still have excessive protein intake. Thus, there should be no problem in further reducing the protein level of formula during the first 6 months of life by increasing the proportion of alpha-lactalbumin. In this way the investigators might achieve a growth pattern and a metabolism more similar to that of the breast-fed infant. Acid whey protein is already in use today by some producers to obtain whey to casein ratio more similar to that of breast milk and to increase the concentration of tryptophan, which is an alternative, in increasing the proportion of alpha-lactalbumin. In this study the investigators intend to study both possibilities.

Alpha-lactalbumin has been suggested to influence the gut bacterial flora with a positive antimicrobial effect and improved immune function of the infant. Hypothetically, an increased intake of alpha-lactalbumin may result in fewer infections in formula-fed infants and thus decrease the differences in infection prevalence between formula- and breast-fed infants. Alpha-lactalbumin also seems to influence the uptake of minerals, such as iron, which could be important for iron status of the infant. Thus, iron status may improve in formula-fed infants when alpha-lactalbumin is added to formula, which has previously been shown by us and others.

With metabolomics, chemical processes involving metabolites, small molecule substrates, intermediates and products of metabolism are studied. Specifically, metabolomics is identifies a unique chemical fingerprints that specific cellular processes leave behind". Differences in metabolomics between the different groups will be studied Objectives: The purpose of the present study is to evaluate the effect of feeding infants a protein-reduced infant formula with high or low levels of alpha-lactalbumin on growth, metabolic markers and gut microbiota composition.

Methods: Healthy infants with normal growth parameters will be included. If the infant is fully formula-fed at 4-8 weeks of age, he or she will be randomized in a double blinded controlled manner to one of the three formula groups and receive the assigned infant formula until 6 month of age. The investigators will also include exclusively breast fed infants, whose mothers intend to breast-feed for at least 6 months, in a breastfed group.

From inclusion through the 12th month of age dietary intake, the incidence and duration of illness, stool consistency, fever, gastrointestinal problems, respiratory problems, and during the first 6 months also sleep- and crying time, will be recorded by the parents. Hospitalization and unscheduled doctor's visits will also be recorded by parents as well as medication (type, duration) and any adverse effects. Growth and well-being will be followed. Blood samples will be taken for analyses of protein metabolism and metabolomics and fecal microbiota will be analyzed as well as metabolites in urine.

Outcomes: Through this study the investigators should be able to clarify if feeding infants a protein-reduced formula with addition of alpha-lactalbumin or acid whey protein will affect growth, metabolic markers, gut microbiota composition and health parameters to approach those of breast-fed infants with possibly lower risk of overweight in childhood and lower incidences of infections in formula-fed infants.

ELIGIBILITY:
Inclusion

* Healthy infants
* Born vaginally (no caecerian section)
* 37+0 until 42+0
* Birth weight ± 2 SD of internationally approved growth charts
* No severe neonatal problems
* No feeding problems
* No evidence of systemic disease

Exclusion Criteria:

* Partial breast feeding at 8 weeks
* Breast feeding in the formula Group
* Formula feeding in the breast fed Group
* Caecerian section
* Treatment with antibiotics during the first 8 weeks

Ages: 4 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 328 (Actual)
Dates: Start 2014-11; Primary Completion 2020-04 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Growth | 5 years
  body composition

SECONDARY OUTCOMES:
Gut microbiota | 5 years
  Feacal tests
Infection frequency | 1 year
  Reported infections
sleep | 2-6 months
  sleep latency

CONTACTS AND LOCATIONS:
Overall Officials: Pia M Karlsland Åkeson, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lonnerdal B, Lien EL. Nutritional and physiologic significance of alpha-lactalbumin in infants. Nutr Rev. 2003 Sep;61(9):295-305. doi: 10.1301/nr.2003.sept.295-305. PMID 14552064
- [Background] ESPGHAN Committee on Nutrition; Agostoni C, Braegger C, Decsi T, Kolacek S, Koletzko B, Michaelsen KF, Mihatsch W, Moreno LA, Puntis J, Shamir R, Szajewska H, Turck D, van Goudoever J. Breast-feeding: A commentary by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2009 Jul;49(1):112-25. doi: 10.1097/MPG.0b013e31819f1e05. PMID 19502997
- [Background] Karlsland Akeson PM, Axelsson IE, Raiha NC. Protein and amino acid metabolism in three- to twelve-month-old infants fed human milk or formulas with varying protein concentrations. J Pediatr Gastroenterol Nutr. 1998 Mar;26(3):297-304. doi: 10.1097/00005176-199803000-00011. PMID 9523865
- [Background] Axelsson IE, Jakobsson I, Raiha NC. Formula with reduced protein content: effects on growth and protein metabolism during weaning. Pediatr Res. 1988 Sep;24(3):297-301. doi: 10.1203/00006450-198809000-00004. PMID 3062558
- [Derived] He X, Tinghall Nilsson U, Mishchuk DO, Hernell O, Lonnerdal B, Hartvigsen ML, Jacobsen LN, Kvistgaard AS, Slupsky CM, Karlsland Akeson P. Impact of formula protein quantity and source on infant metabolism: serum, urine, and fecal metabolomes of a randomized controlled study. Am J Clin Nutr. 2025 Apr;121(4):853-864. doi: 10.1016/j.ajcnut.2025.02.002. Epub 2025 Feb 5. PMID 39921093
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765